CLINICAL TRIAL: NCT05492227
Title: SARS-CoV-2 Nucleic Acid Detection Kit
Brief Title: SARS-CoV-2 Nucleic Acid Detection Kit Clinical Performance Study
Acronym: CPS CW008
Status: Completed | Type: Observational
Sponsor: TransGen Biotech Co., LTD (Industry)
Responsible Party: Sponsor
Other Study IDs: CW008
Record Dates: First submitted 2022-08-02; First posted 2022-08-08 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: COVID-19; Coronavirus Disease 2019; COVID-19 Pandemic; Diagnoses Disease
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fresh left-over specimens of SARS-CoV-2 positive subject swabs: All fresh swab specimens that were sent to the biobank Hospital Puerta del Hierro between March 2020 and December 2021 under the standard requirements for SARS-CoV-2 specimens (ISO 201916) were kept frozen (-80ºC) after analysis by RT-PCR (left-over samples).
  Interventions: Diagnostic Test: Left-overs
- Fresh left-over specimens of SARS-CoV-2 negative subject swabs: All fresh swab specimens that were sent to the biobank Hospital Puerta del Hierro between March 2020 and December 2021 under the standard requirements for SARS-CoV-2 specimens (ISO 201916) were kept frozen (-80ºC) after analysis by RT-PCR (left-over samples).
  Interventions: Diagnostic Test: Left-overs

INTERVENTIONS:
Diagnostic Test: Left-overs — Totally nasal swab leftovers were stored from the biobank of Hospital Puerta del Hierro. The coded specimens were kept at -80°C and analyzed using the SARS-CoV-2 NAD Kit. Previously these specimens were analyzed using the gold-standard RT-PCR.

SUMMARY:
SARS-CoV-2 Nucleic Acid Detection Kit is an In Vitro Diagnostic (IVD) medical device intended for RNA detection of SARS-CoV-2 in human specimens using multiplex real-time polymerase chain reaction (RT-PCR) technology. The conserved regions of ORF1ab and N genes are used as target sites of the primers and probes according to the indications provided in the Instructions for Use (IFU).

DETAILED DESCRIPTION:
The SARS-CoV-2 Nucleic Acid Detection Kit is an In Vitro Diagnostic (IVD) medical device intended for Qualitative RNA detection of SARS-CoV-2 using multiplex real time RT-PCR technology for professional use. The kit is available in two different formats (48 tests/kit or 200tests/kit), and it can be stored at -20±5ºC away from light for 12 months. This kit includes a PCR Reaction Mix, PCR Enzyme Mix, SARS-CoV-2 PCR Primer/Probe Mix and a negative/positive control.

TransGen SARS-CoV-2 Nucleic Acid Detection Kit is intended for in vitro qualitative detection of ORF1ab and N genes from the SARS-CoV-2 virus in nasopharyngeal swab specimens collected from COVID-19 suspected cases, suspected clusters of cases or other individuals who need SARS-CoV-2 infection diagnosis or differentiation diagnosis. The definitions of COVID-19-related groups, such as "suspected cases" or "suspected clusters of cases", are detailed in the Diagnosis and Treatment Protocol for Novel Corona virus Pneumonia, Surveillance Protocol for Novel Corona virus Pneumonia or other COVID-19 documents from the Centers for Disease Control and Prevention (CDC). The TransGen SARS-CoV-2 Nucleic Acid Detection Kit should comply with the requirements of Diagnosis and Treatment Protocol for Novel Corona virus Pneumonia, Protocol for Prevention and Control of COVID-19 and other COVID-19 documents from the CDC. The biosafety requirements should be strictly followed as well.

Specimens used for this clinical performance study will be remnants of specimens taken for purposes of standard of care (leftover or archived) through a nasal swab from male and female subjects. Specimens may come from persons suspected of SARS-CoV-2 infection but also from those who need a diagnostic test due to other reasons such as medical intervention, blood donors, or travel for which a negative test is requested.

ELIGIBILITY:
Inclusion Criteria:

* Specimen collected with a nasal swab.
* Negative samples from specimens confirmed SARS-CoV-2 negative by the gold standard, or positive samples from specimens confirmed SARS-CoV-2 positive by the gold standard.

Exclusion Criteria:

* Specimens that have been stored at 4ºC for more than 24h
* Specimens stored at -70ºC that have been under more than 2 freeze/thaw cycles
* Specimens that have been stored at -20 for more than 10 days
* Contamination and/or deterioration of the specimen that, in the investigator's opinion, may impact its handling and/or analysis

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The specimens used in this clinical performance study are leftovers previously collected from male and female subjects suspected of SARS-CoV-2 infection through a nasopharyngeal swab.
Sampling Method: Non-Probability Sample
Enrollment: 607 (Actual)
Dates: Start 2022-07-05 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Sensitivity of the SARS-CoV-2 NAD Kit | Immediately after the procedure
  The investigators assessed the sensitivity as the capacity to correctly detect positive specimens of SARS-CoV-2 infection previously confirmed as positive (True Positive, TP) by the gold standard RT-PCR.

SECONDARY OUTCOMES:
Specificity of the SARS-CoV-2 NAD Kit | Immediately after the procedure
  The investigators assessed the specificity as the ability to correctly classify previously confirmed as SARS-CoV-2 negative specimens by the gold standard RT-PCR, as negative (True Negative, TN).

CONTACTS AND LOCATIONS:
Locations (1):
- Biobanco del Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No